CLINICAL TRIAL: NCT02551458
Title: SYSTEMATIC SURGERY VERSUS SURVEILLANCE AND RESCUE SURGERY IN OPERABLE CANCER OF THE OESOPHAGUS WITH A COMPLETE CLINICAL RESPONSE TO RADIOCHEMOTHERAPY
Brief Title: Comparison of Systematic Surgery Versus Surveillance and Rescue Surgery in Operable Oesophageal Cancer With a Complete Clinical Response to Radiochemotherapy
Acronym: Esostrate
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: sub-optimal inclusion rate, additional 9 years to finalize inclusion and follow-up of all patients.
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Bedenne PHRC N 2013
Record Dates: First submitted 2015-08-20; First posted 2015-09-16 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Epidermoid Carcinoma or; Adenocarcinoma of the Thoracic Oesophagus or; Adenocarcinoma of the Oesogastric Junction (Siewert Type I or II); Stage cT2 N1-3 M0 or cT3-T4a N0 or N1-3 M0
MeSH Terms: conditions — Carcinoma, Squamous Cell

ARMS (2):
- Arm A: Systematic surgery (Experimental)
  Interventions: Other: Systematic surgery
- Arm B: Surveillance and rescue surgery in cases of resectable (Experimental)
  Interventions: Other: Surveillance and rescue surgery in cases of resectable loco-regional recurrence

INTERVENTIONS:
Other: Systematic surgery
  Arms: Arm A: Systematic surgery
Other: Surveillance and rescue surgery in cases of resectable loco-regional recurrence
  Arms: Arm B: Surveillance and rescue surgery in cases of resectable

SUMMARY:
Step 1: Inclusion of eligible patients to carry out a translational search for prognostic and predictive markers of Complete Clinical Response and Pathologic Complete Response (using blood samples and diagnostic biopsies) and to collect data on radiochemotherapy and its toxicity.

The trial will evaluate strategies after neoadjuvant treatment and not RCT protocols. The RCT will thus be chosen by the investigator from published effective schemes in a pre-operative setting or in patients not undergoing surgery.

Evaluation of the response 5 to 6 weeks after the RCT.

Step 2: Randomisation in patients with a complete clinical response:

Arm A: Systematic surgery Arm B: Surveillance and rescue surgery in cases with resectable loco-regional recurrence

Patients not eligible for randomisation will have the possibility to participate in a specific study (information can be obtained from the SAKK group (Switzerland Group Clinical Research on Cancer)).

ELIGIBILITY:
Inclusion Criteria:

* Epidermoid carcinoma (EC) or adenocarcinoma of the thoracic oesophagus or adenocarcinoma of the oesogastric junction (Siewert type I or II) proven histologically
* Stage cT2 N1-3 M0 or cT3-T4a N0 or N1-3 M0 after a full investigation
* Patient considered operable with a curative intent and scheduled to undergo first-line radiochemotherapy in a multidisciplinary meeting
* Age ≥ 18 years < 75 years
* Patient with national health insurance cover and who has provided written informed consent for the clinical and biological studies.

Exclusion Criteria:

* Cancer of the cervical oesophagus (15 to 19 cm from the dental arches)
* Weight loss > 15% at the recruitment with no improvement after nutritional support
* Serious comorbidity threatening survival in the short term
* Contra-indication for radiochemotherapy
* Other uncured malignant disease in the 5 previous years (except for in situ cervical carcinoma and treated non-melanotic skin cancers)
* Absence of effective contraception in patients (men or women) able to procreate, pregnant or breast-feeding women
* Impossibility to follow the trial
* Legal disqualification (patients in custody or under guardianship)

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Proportion of surviving patients | 1 year after randomisation
Disease-free survival | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - CHU Amiens, Amiens
  - Centre d'oncologie et de radiothérapie du Pays Basque, Bayonne
  - CH de la Côte Basque, Bayonne
  - Boulogne Sur Mer, Boulogne-sur-Mer
  - Infirmerie protestante de Lyon, Caluire-et-Cuire
  - Hôpitaux civils de Colmar, Colmar
  - CHU de DIJON, Dijon
  - Hôpital Michallon (GRENOBLE), La Tronche
  - Centre Oscar Lambret, Lille
  - Hôpital Claude Huriez, Lille
  - Clinique Chenieux, Limoges
  - CHU de Limoges, Limoges
  - CH Saint Joseph Saint Luc, Lyon
  - Hôpital privé Jean Mermoz, Lyon
  - Institut Mutualiste MONTSOURIS, Paris
  - Centre Hospitalier Annecy Genevois, Pringy
  - CHP Saint Grégoire, Saint-Grégoire
  - Institut Gustave Roussy, Villejuif